CLINICAL TRIAL: NCT05343871
Title: Randomized Controlled Trial to Assess the Immunogenicity and Safety of Full Versus Fractional Dose of Pfizer/BioNTech, AstraZeneca, and Sinovac COVID-19 Vaccines Given as a Booster Dose at Least 6 Months After Primary Vaccination Series or PCR-confirmed Infection With SARS-CoV-2 in Healthy Adults
Brief Title: Immunogenicity and Safety of Fractional Booster Dose of COVID-19 Vaccines Available for Use in Pakistan/Brazil: A Phase 4 Dose-optimizing Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Collaborators: Aga Khan University (Other); Oswaldo Cruz Foundation (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sabin CoV 22
Record Dates: First submitted 2022-04-20; First posted 2022-04-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: Fractional dose; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; ChAdOx1 nCoV-19; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be observer-blind. Participants, data collectors (e.g., Investigator), and data evaluators (e.g., trial statisticians) are blinded. Only the staff involved in vaccine delivery will be unblinded and aware of which vaccine the participant is receiving (group allocation). Study staff who collect information on symptoms and adverse events, laboratory staff and statisticians conducting the analysis will all be blinded to the vaccine and dosage received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (19):
- Priming Group 1: Sinovac Prime, AZD1222 ½ dose (Brazil only) (Experimental)
  Interventions: Biological: AZD1222
- Priming Group 1: Sinovac Prime, AZD1222 full dose (Brazil only) (Active Comparator)
  Interventions: Biological: AZD1222
- Priming Group 1: Sinovac Prime, BNT162b2 1/3 dose (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 1: Sinovac Prime, BNT162b2 1/2 dose (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 1: Sinovac Prime, BNT162b2 full dose (Active Comparator)
  Interventions: Biological: BNT162b2
- Priming Group 1: Sinovac Prime, Sinovac full dose (Active Comparator)
  Interventions: Biological: Sinovac
- Priming Group 2: AZD1222 Prime, AZD1222 ½ dose (Brazil only) (Experimental)
  Interventions: Biological: AZD1222
- Priming Group 2: AZD1222 Prime, AZD1222 full dose (Brazil only) (Active Comparator)
  Interventions: Biological: AZD1222
- Priming Group 2: AZD1222 Prime, BNT162b2 1/3 dose (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 2: AZD1222 Prime, BNT162b2 1/2 dose (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 2: AZD1222 Prime, BNT162b2 full dose (Active Comparator)
  Interventions: Biological: BNT162b2
- Priming Group 3-B: BNT162b2 Prime, AZD1222 ½ dose (Brazil only) (Experimental)
  Interventions: Biological: AZD1222
- Priming Group 3-B: BNT162b2 Prime, AZD1222 full dose (Brazil only) (Active Comparator)
  Interventions: Biological: AZD1222
- Priming Group 3-B: BNT162b2 Prime, BNT162b2 1/3 dose (Brazil only) (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 3-B: BNT162b2 Prime, BNT162b2 1/2 dose (Brazil only) (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 3-B: BNT162b2 Prime, BNT162b2 full dose (Brazil only) (Active Comparator)
  Interventions: Biological: BNT162b2
- Priming Group 3-P: Natural Infection Prime, BNT162b2 1/3 dose (Pakistan only) (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 3-P: Natural Infection Prime, BNT162b2 1/2 dose (Pakistan only) (Experimental)
  Interventions: Biological: BNT162b2
- Priming Group 3-P: Natural Infection Prime, BNT162b2 full dose (Pakistan only) (Active Comparator)
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: Sinovac — Sinovac inactivated COVID-19 vaccine:
  ● Full dose (0.5 ml)
  Arms: Priming Group 1: Sinovac Prime, Sinovac full dose
Biological: AZD1222 — AstraZeneca ChAdOx1-S recombinant AZD1222 vaccine:
  * Full dose (0.5 ml)
  * Half dose (0.25 ml)
  Arms: Priming Group 1: Sinovac Prime, AZD1222 full dose (Brazil only); Priming Group 1: Sinovac Prime, AZD1222 ½ dose (Brazil only); Priming Group 2: AZD1222 Prime, AZD1222 full dose (Brazil only); Priming Group 2: AZD1222 Prime, AZD1222 ½ dose (Brazil only); Priming Group 3-B: BNT162b2 Prime, AZD1222 full dose (Brazil only); Priming Group 3-B: BNT162b2 Prime, AZD1222 ½ dose (Brazil only)
Biological: BNT162b2 — Pfizer/BioNTech BNT162b2 mRNA vaccine:
  * Full dose (30 micrograms)
  * Half dose (15 micrograms)
  * One-third dose (10 micrograms)
  Arms: Priming Group 1: Sinovac Prime, BNT162b2 1/2 dose; Priming Group 1: Sinovac Prime, BNT162b2 1/3 dose; Priming Group 1: Sinovac Prime, BNT162b2 full dose; Priming Group 2: AZD1222 Prime, BNT162b2 1/2 dose; Priming Group 2: AZD1222 Prime, BNT162b2 1/3 dose; Priming Group 2: AZD1222 Prime, BNT162b2 full dose; Priming Group 3-B: BNT162b2 Prime, BNT162b2 1/2 dose (Brazil only); Priming Group 3-B: BNT162b2 Prime, BNT162b2 1/3 dose (Brazil only); Priming Group 3-B: BNT162b2 Prime, BNT162b2 full dose (Brazil only); Priming Group 3-P: Natural Infection Prime, BNT162b2 1/2 dose (Pakistan only); Priming Group 3-P: Natural Infection Prime, BNT162b2 1/3 dose (Pakistan only); Priming Group 3-P: Natural Infection Prime, BNT162b2 full dose (Pakistan only)

SUMMARY:
Since the emergence of the novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pathogen in late 2019, millions of people around the world have fallen ill and died from coronavirus disease 2019 (COVID-19), with variant-fueled case spikes causing repeated cycles of morbidity and mortality. The rapid development and emergency use authorization of vaccines against SARS-CoV-2 presents an enormous opportunity to protect populations, but bottlenecks in production have led to demand for vaccines that far outpaces supply. This project will investigate the immunogenicity of fractional doses of SARS-CoV-2 vaccines given a minimum of six months following an initial two-dose schedule or following natural immunity via documented infection. The consortium of research partners from the Sabin Vaccine Institute, Aga Khan University, Fundação Oswaldo Cruz (Fiocruz), and Stanford University will recruit volunteers to receive a full or fractional booster dose of BNT162b2, AZD1222 or Sinovac following receipt of their primary vaccination series or PCR-confirmed natural infection in Pakistan. The research team will follow participants for six months from boosting, with blood draws at baseline, 28 days, 3 months and 6 months, and measure sero-response rate (SRR) by anti-Spike immunoglobulin G (IgG) binding enzyme-linked immunosorbent assay (ELISA) with the ultimate aim of identifying whether fractional doses provide a similar immune response compared to full doses of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female individuals aged 18 years to 60 years
* Participant is willing and able to give written informed consent for participation in the trial
* Individuals who can comply with trial procedures and are available for the duration of follow-up.

Brazil:

● Previous vaccination with a complete primary series of Sinovac (Priming Group 1), AZD1222 (Priming Group 2), or BNT162b2 (Priming Group 3-B) at least 6 months prior to screening

Pakistan:

● Previous vaccination with a complete primary series of Sinovac (Priming Group 1) or AZD1222 (Priming Group 2) at least 6 months prior to screening, or PCR-confirmed natural infection (Priming Group 3-P) between February 2021 - 6 months prior to screening

Exclusion Criteria:

* Has a contraindication to BNT162b2, AZD1222 or Sinovac
* Has received an incomplete primary COVID-19 vaccination series
* Has received 3 doses of COVID-19 vaccine
* Has received heterologous primary COVID-19 vaccination series
* History of a solid organ or bone marrow transplant
* History of malignancy (other than non-melanoma skin cancer) within the past five years
* Currently on hemodialysis
* Any confirmed or suspected immunosuppressive or immunodeficiency condition or diagnosis
* On chronic (>30 days) use of immunosuppressive medications at the time of enrollment (except topical steroids or short-term oral steroids, i.e., ≤14 days)
* Known diagnosis of HIV with CD4 count <200 cells/mm3 (in the past 6 months)
* Active or history of previous auto-immune neurological disorders (e.g., multiple sclerosis, Guillain-Barre syndrome, transverse myelitis) (excluding Bell's palsy)
* Has received anti-CD20 monoclonal antibodies for any reason in the past 12 months
* Has received monoclonal antibodies to treat a previous COVID-19 event
* Pregnant at screening
* Positive SARS-CoV-2 Antigen test in respiratory specimen at screening
* Planning to migrate out of the study area within 6 months of the enrollment
* Participants currently enrolled in any other COVID-19 vaccine research trial in which they are getting a COVID-19 vaccine during the study period
* Illiterate individuals (Brazil only)
* Has a severe and/or uncontrolled comorbidity

Pakistan (natural infection Priming Group (Priming Group 3-P)):

● Prior vaccination with ANY vaccine against COVID-19

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2354 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Sero-response rate by Spike IgG binding ELISA at 28 days post booster | Day 28
  Assess and compare humoral immune response from a fractional vs. full booster dose of BNT162b2 or AZD1222 in immunocompetent adults fully primed with BNT162b2, AZD1222, or Sinovac vaccines or natural infection, measured by anti-Spike IgG binding ELISA at 28 days post booster
Safety and reactogenicity profile of fractional and full dose of study vaccines at 28 days post-booster vaccination | Day 28
  Describe the safety and reactogenicity profile of fractional and full dose of study vaccines at 28 days post-booster vaccination through estimated incidence of solicited local and systemic adverse events, and incidence of unsolicited reported adverse events
  1. Occurrence of solicited local and systemic reactions within 7 days of booster
  2. Occurrence of unsolicited AEs within 28 days of booster

SECONDARY OUTCOMES:
Sero-response rate by anti-Spike IgG binding ELISA at 3m and 6m post booster | Month 3 and Month 6
  Assess the persistence of humoral immunity after a fractional vs. full booster dose of BNT162b2 or AZD1222 in immunocompetent adults fully primed with BNT162b2, AZD1222, or Sinovac vaccines or natural infection, measured by anti-Spike IgG binding ELISA at 3m and 6m post booster
Safety and reactogenicity profile of fractional and full dose of study vaccines throughout the trial | Throughout study, 6 months per participant
  Describe the safety and reactogenicity profile of fractional and full dose of study vaccines throughout the trial
  1. Occurrence of Medically attended adverse reactions within 3 months of booster
  2. Occurrence of adverse events (AE), Serious adverse events (SAE), and adverse events of special interest (AESI) within 28 days, 3 months, and 6 months of booster

CONTACTS AND LOCATIONS:
Locations (2):
- FIOCRUZ, Campo Grande, MS Do Sul, Brazil
- Aga Khan University Clinical Trials Unit, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Barros Verruck J, Moreira Puga MA, de Oliveira RD, Vieira da Silva P, Charu V, Hedlin H, Lu D, Zhang A, Ritter V, Shaw B, Rosser JI, Seidman JC, Carter AS, Qamar F, Luby S, Garret D, Croda J. Antispike IgG antibody decay after immunisation with fractional versus full booster doses of COVID-19 vaccines: a 6-month longitudinal analysis of the FRACT-COV trial in Brazil. BMJ Public Health. 2025 Jul 5;3(2):e002331. doi: 10.1136/bmjph-2024-002331. eCollection 2025. PMID 40620571